CLINICAL TRIAL: NCT01115855
Title: The Effect Of Eplerenone Versus Placebo On Cardiovascular Mortality And Heart Failure Hospitalization In Japanese Subjects With Chronic Heart Failure
Brief Title: Clinical Study Of Eplerenone In Japanese Patients With Chronic Heart Failure
Acronym: J-EMPHASIS-HF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A6141114
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Results first posted 2016-10-27 (Estimated); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Heart Failure
Keywords: Double-blind; eplerenone; Japanese
MeSH Terms: conditions — Heart Failure | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eplerenone arm (Experimental): Add on standard heart failure therapy
  Interventions: Drug: Eplerenone
- Placebo arm (Placebo Comparator): Add on standard heart failure therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eplerenone — Eplerenone 25 mg once every other day, 25mg once daily or 50 mg once daily
  Arms: Eplerenone arm
Drug: Placebo — Placebo once daily or every once daily
  Arms: Placebo arm

SUMMARY:
A study to compare the efficacy and safety of eplerenone in Japanese chronic heart failure patients with placebo.

DETAILED DESCRIPTION:
The aim of this study was to show consistency with the EMPHASIS-HF trial (NCT00232180), which was defined as a HR of the primary endpoint of below 1.

ELIGIBILITY:
Inclusion Criteria:

* Japanese chronic systolic heart failure patients with LVEF =<30% by echocardiography and NYHA II or more
* Patients who receive standard therapy (Angiotensin converting enzyme inhibitors, angiotensin receptor blockers, beta-blocker or diuretic)

Exclusion Criteria:

* Patients with a myocardial infarction, stroke, cardiac surgery or percutaneous coronary intervention within 30 days prior to randomization.
* Patients with serum potassium >5.0 mmol/L or eGFR <30 ml/min/1.73 m2.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2010-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (54):
- Japan (54):
  - Chubu Rosai Hospital, Nagoya, Aichi-ken
  - Tosei General Hospital, Seto, Aichi-ken
  - Asahi General Hospital, Asahi, Chiba
  - National Hospital Organization Chiba Medical Center, Chiba, Chiba
  - Nippon Medical School Chiba Hokusou Hospital, Inzai, Chiba
  - Ehime Prefectural Central Hospital, Matuyama-shi, Ehime
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Aso Iizuka Hospital, Iizuka-shi, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Southern TOHOKU Research Institute for Neuroscience Southern TOHOKU Medical Clinic, Kōriyama, Fukushima
  - Ogaki Municipal Hospital, Ōgaki, Gifu
  - National Hospital Organization Hakodate National Hospital, Hakodate-shi, Hokkai-do
  - Hakodate City Hospital, Hakodate, Hokkaido
  - Teine Keijinkai Clinic, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - National Hospital Organization Hokkaido Medical Center, Sapporo, Hokkaido
  - Hyogo Brain and Heart Center, Himeji, Hyōgo
  - Japanease Red Cross Society Himeji Hospital, Himeji, Hyōgo
  - The Hospital of Hyogo College of Medicine, Nishinomiya, Hyōgo
  - Toride Kyodo General Hospital, Toride-shi, Ibaraki
  - Mitoyo General Hospital, Kan’onjichō, Kagawa-ken
  - Fujisawa City Hospital, Fujisawa, Kanagawa
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Mie University Hospital, Tsu, Mie-ken
  - National Hospital Organization Sendai Medical Center, Sendai, Miyagi
  - Nara Medical University Hospital, Kashihara, Nara
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - Sakai City Medical Center, Sakai-shi, Osaka
  - National Cerebral and Cardiovascular Center Hospital, Suita-shi, Osaka
  - Gokeikai Osaka Kaisei Hospital, Yodogawa-ku, Osaka
  - Shuwa General Hospital, Kasukabe-shi, Saitama
  - Saitama Medical Center Jichi Medical University, Saitama-shi, Saitama
  - Kusatsu General Hospital, Kusatsu-shi, Shiga
  - Hamamatsu Rosai Hospital, Hamamatsu, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke-shi, Tochigi
  - Tokushima Red Cross Hospital, Komatsushimachō, Tokushima
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Mitsui Memorial Hospital, Chiyoda-Ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Tottori University Hospital, Yonago-shi, Tottori
  - Ube-kohsan Central Hospital Corp., Ube, Yamaguchi
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - University of Yamanashi Hospital, Chūō, Yamanashi
  - Hamanomachi Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Gifu Prefectural General Medical Center, Gifu
  - Kumamoto University Hospital, Kumamoto
  - Saiseikai Kumamoto Hospital, Kumamoto
  - Japanese Red Cross Okayama Hospital, Okayama
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka Police Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - National Hospital Organization Takasaki General Medical Center, Takasaki-shi
  - Toyama University Hospital, Toyama

REFERENCES:
- [Derived] Tsutsui H, Ito H, Kitakaze M, Komuro I, Murohara T, Izumi T, Sunagawa K, Yasumura Y, Yano M, Yamamoto K, Yoshikawa T, Tsutamoto T, Zhang J, Okayama A, Ichikawa Y, Kanmuri K, Matsuzaki M; J-EMPHASIS-HF Study Group. Double-Blind, Randomized, Placebo-Controlled Trial Evaluating the Efficacy and Safety of Eplerenone in Japanese Patients With Chronic Heart Failure (J-EMPHASIS-HF). Circ J. 2017 Dec 25;82(1):148-158. doi: 10.1253/circj.CJ-17-0323. Epub 2017 Aug 19. PMID 28824029

RESULTS

PARTICIPANT FLOW:
Groups:
- Eplerenone: Participants with estimated glomerular filtration rate (eGFR) greater than or equal to (>=) 50 milliliter per minute divided by 1.73 squared meter (mL/min/1.73m^2) received eplerenone 25 milligram (mg) tablet once daily up to Week 4 and participants with eGFR 30 to less than (<) 50 mL/min/1.73m^2 received eplerenone 25 mg tablet every other day up to Week 4. . From Week 4 onward, the dose of eplerenone was limited to 50 mg once daily for participants with eGFR >=50 mL/min/1.73 m^2 and 25 mg once daily for participants with eGFR 30 to <50 mL/min/1.73 m^2 up to Month 48.
- Placebo: Participants with eGFR >=50 mL/min/1.73m^2 received placebo matched with eplerenone tablet orally once daily from up to Week 4 and participants with eGFR 30 to <50 mL/min/1.73m^2 received placebo matched with eplerenone tablet every other day up to Week 4. From Week 4 onward, all participants received placebo matched with eplerenone tablet once daily up to Month 48.
Period: Overall Study
Arm/Group | Eplerenone | Placebo
Started | 111 | 110
Completed | 75 | 74
Not Completed | 36 | 36
Not completed — Adverse Event | 16 | 18
Not completed — Death | 6 | 5
Not completed — Lab Abnormality | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Other | 8 | 6

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomized participants.
Groups:
- Eplerenone: Participants with eGFR >=50 mL/min/1.73m^2 received eplerenone 25 mg tablet once daily up to Week 4 and participants with eGFR 30 to < 50 mL/min/1.73m^2 received eplerenone 25 mg tablet every other day up to Week 4. From Week 4 onward, the dose of eplerenone was limited to 50 mg once daily for participants with eGFR >=50 mL/min/1.73 m^2 and 25 mg once daily for participants with eGFR 30 to <50 mL/min/1.73 m^2 up to Month 48.
- Total: Total of all reporting groups
Arm/Group | Eplerenone | Placebo | Total
Number analyzed (Participants) | 111 | 110 | 221
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (8.7) | 68.4 (7.7) | 68.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  FEMALE | 26 | 19 | 45
  MALE | 85 | 91 | 176

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Occurrence of Cardiovascular (CV) Mortality or Hospitalization Due to Heart Failure (HF)
Description: CV mortality was defined as any death due to HF, myocardial infarction, cardiac arrhythmia, stroke or cerebral vascular accident, other CV cause (such as aneurysm or pulmonary embolism). Hospitalization due to HF was defined as an overnight stay, or longer, in a hospital environment (emergency room, observation unit or in-patient care, or similar facility including admission to a day care facility) due to HF. Hazard ratio of Eplerenone versus placebo for first occurrence of the event was obtained from a Cox proportional hazards model.
Time Frame: Randomization up to the date when the last enrolled participant had been followed up for 1 year (up to 1744 days)
Population: Full analysis set included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 111 | 110
participants | 33 | 36
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; Cox Proportional Hazard Model with baseline New York Heart Association (NYHA) cohort (II, III/IV) and baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) covariates; Test type: Superiority or Other; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.53 to 1.36]

2. Secondary Outcome: Number of Participants With First Occurrence of Cardiovascular (CV) Mortality, Hospitalization Due to Heart Failure (HF), or Addition/Increase of Heart Failure (HF) Medication
Description: CV mortality was defined as any death due to HF, myocardial infarction, cardiac arrhythmia, stroke or cerebral vascular accident, other CV cause (such as aneurysm or pulmonary embolism). Hospitalization due to HF was defined as an overnight stay, or longer, in a hospital environment (emergency room, observation unit or in-patient care, or similar facility including admission to a day care facility) due to HF. Addition/ increase of HF medications was defined as administration of new HF medication or increase of 50 percentage (%) or more in dose of HF medication for >= 3 days. Hazard ratio of Eplerenone versus placebo for first occurrence of the event was obtained from a Cox proportional hazards model.
Time Frame: Randomization up to the date when the last enrolled participant had been followed up for 1 year (up to 1744 days)
Population: Full analysis set included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 111 | 110
participants | 42 | 45
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; Cox Proportional Hazard Model with baseline NYHA cohort (II, III/IV) and baseline eGFR (30--<50 ml/min/1.73 m^2, >-=50 ml/min/1.73 m^2) covariates; Test type: Superiority or Other; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.56 to 1.31]

3. Secondary Outcome: Number of Participants With With First Occurrence of All-Cause Mortality
Description: All-cause mortality was defined as any CV mortality, Non-CV mortality, including malignant tumor, pulmonary disease and trauma.CV mortality was defined as death due to HF, myocardial infarction, cardiac arrhythmia, stroke or cerebral vascular accident, other CV cause (such as aneurysm or pulmonary embolism). Mortality during treatment, within 30 days of treatment discontinuation and after 30 days of discontinuation was reported. Hazard ratio of Eplerenone versus placebo for first occurrence of the event was obtained from a Cox proportional hazards model.
Time Frame: Randomization up to the date when the last enrolled participant had been followed up for 1 year (up to 1744 days)
Population: Full analysis set included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 111 | 110
participants
  During treatment | 6 | 5
  Within 30 days of treatment discontinuation | 1 | 1
  After 30 days of treatment discontinuation | 10 | 4
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 1.77, 95% CI 2-sided [0.81 to 3.87]

4. Secondary Outcome: Number of Participants With With First Occurrence of Cardiovascular Mortality
Description: CV mortality was defined as death due to HF, myocardial infarction, cardiac arrhythmia, stroke or cerebral vascular accident, other CV cause (such as aneurysm or pulmonary embolism). Hazard ratio of Eplerenone versus placebo for first occurrence of the event was obtained from a Cox proportional hazards model.
Time Frame: Randomization up to the date when the last enrolled participant had been followed up for 1 year (up to 1744 days)
Population: Full analysis set included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 111 | 110
participants | 14 | 6
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 2.40, 95% CI 2-sided [0.92 to 6.24]

5. Secondary Outcome: Number of Participants With First Occurrence of All-cause Hospitalization
Description: All cause hospitalization included all hospitalizations as CV hospitalization, which was defined as any hospitalization due to CV events including HF, myocardial infarction, arrhythmia, angina pectoris and non-CV hospitalizations which was defined as any hospitalization due to non-CV events including renal dysfunction, hyperkalaemia, malignant tumor and pulmonary disease. Hazard ratio of Eplerenone versus placebo for first occurrence of the event was obtained from a Cox proportional hazards model.
Time Frame: Randomization up to the date when the last enrolled participant had been followed up for 1 year (up to 1744 days)
Population: Full analysis set included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 111 | 110
participants | 45 | 58
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.44 to 0.97]

6. Secondary Outcome: Number of Participants With First Occurrence of Hospitalization Due to Heart Failure (HF)
Description: Hospitalization due to HF was defined as an overnight stay, or longer, in a hospital environment (emergency room, observation unit or in-patient care, or similar facility including admission to a day care facility) due to HF. Hazard ratio of Eplerenone versus placebo for first occurrence of the event was obtained from a Cox proportional hazards model.
Time Frame: Randomization up to the date when the last enrolled participant had been followed up for 1 year (up to 1744 days)
Population: Full analysis set included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 111 | 110
participants | 27 | 33
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.45 to 1.25]

7. Secondary Outcome: Number of Participants With First Occurrence of All-cause Mortality or All-cause Hospitalization
Description: All cause hospitalization included all hospitalizations as CV hospitalization, which was defined as any hospitalization due to CV events including HF, myocardial infarction, arrhythmia, angina pectoris and non-CV hospitalizations which was defined as any hospitalization due to non-CV events including renal dysfunction, hyperkalaemia, malignant tumor and pulmonary disease. All-cause mortality was defined as any CV mortality, Non-CV mortality, including malignant tumor, pulmonary disease and trauma.CV mortality was defined as death due to HF, myocardial infarction, cardiac arrhythmia, stroke or cerebral vascular accident, other CV cause (such as aneurysm or pulmonary embolism). Hazard ratio of Eplerenone versus placebo for first occurrence of the event was obtained from a Cox proportional hazards model.
Time Frame: Randomization up to the date when the last enrolled participant had been followed up for 1 year (up to 1744 days)
Population: Full analysis set included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 111 | 110
participants | 48 | 61
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.45 to 0.97]

8. Secondary Outcome: Number of Participants With First Occurrence of Heart Failure (HF) Mortality or Heart Failure (HF) Hospitalization
Description: HF mortality was defined as any death due to HF. Hospitalization due to HF was defined as an overnight stay, or longer, in a hospital environment (emergency room, observation unit or in-patient care, or similar facility including admission to a day care facility) due to HF. Hazard ratio of Eplerenone versus placebo for first occurrence of the event was obtained from a Cox proportional hazards model.
Time Frame: Randomization up to the date when the last enrolled participant had been followed up for 1 year (up to 1744 days)
Population: Full analysis set included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 111 | 110
participants | 29 | 33
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; Cox Proportional Hazard Model with baseline NYHA cohort (II, III/IV) and baseline eGFR (30--<50 ml/min/1.73 m^2, >=-50 ml/min/1.73 m^2) covariates; Test type: Superiority or Other; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.49 to 1.33]

9. Secondary Outcome: Number of Participants With First Occurrence of Cardiovascular (CV) Hospitalization
Description: CV hospitalization, which was defined as any hospitalization due to CV events including HF, myocardial infarction, arrhythmia, angina pectoris. Hazard ratio of Eplerenone versus placebo for first occurrence of the event was obtained from a Cox proportional hazards model.
Time Frame: Randomization up to the date when the last enrolled participant had been followed up for 1 year (up to 1744 days)
Population: Full analysis set included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 111 | 110
participants | 35 | 44
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.45 to 1.10]

10. Secondary Outcome: Number of Participants With First Occurrence of Addition/Increase of Heart Failure (HF) Medication Due to Heart Failure (HF) Worsening
Description: Addition/ increase of HF medications was defined as administration of new HF medication or increase of 50 percent or more in dose of HF medication for >= 3 days. Hazard ratio of Eplerenone versus placebo for first occurrence of the event was obtained from a Cox proportional hazards model.
Time Frame: Randomization up to the date when the last enrolled participant had been followed up for 1 year (up to 1744 days)
Population: Full analysis set included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 111 | 110
participants | 38 | 43
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.53 to 1.28]

11. Secondary Outcome: Number of Participants With First Occurrence of Fatal/Non-Fatal Stroke
Description: Hazard ratio of Eplerenone versus placebo for first occurrence of the event was obtained from a Cox proportional hazards model.
Time Frame: Randomization up to the date when the last enrolled participant had been followed up for 1 year (up to 1744 days)
Population: Full analysis set included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 111 | 110
participants | 3 | 4
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.18 to 3.53]

12. Secondary Outcome: Number of Participants With First Occurrence of Fatal/Non-Fatal Myocardial Infarction (MI)
Description: as for outcome 11
Time Frame: Randomization up to the date when the last enrolled participant had been followed up for 1 year (up to 1744 days)
Population: Full analysis set included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 111 | 110
participants | 1 | 1
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.07 to 17.85]

13. Secondary Outcome: Number of Participants With First Occurrence of New Onset Atrial Fibrillation/Flutter
Description: New onset of atrial fibrillation or flutter was defined as the diagnosis of atrial fibrillation or flutter in a participant after randomization. Hazard ratio of Eplerenone versus placebo for first occurrence of the event was obtained from a Cox proportional hazards model.
Time Frame: Randomization up to the date when the last enrolled participant had been followed up for 1 year (up to 1744 days)
Population: Full analysis set included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 111 | 110
participants | 4 | 2
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 2.11, 95% CI 2-sided [0.39 to 11.56]

14. Secondary Outcome: Number of Participants With First Occurrence of New Onset Diabetes Mellitus
Description: New onset diabetes mellitus was defined as the diagnosis of diabetes mellitus in a participant after randomization. Hazard ratio of Eplerenone versus placebo for first occurrence of the event was obtained from a Cox proportional hazards model.
Time Frame: Randomization up to the date when the last enrolled participant had been followed up for 1 year (up to 1744 days)
Population: Full analysis set included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 111 | 110
participants | 1 | 2
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.05 to 5.66]

15. Secondary Outcome: Number of Participants With First Occurrence of Hospitalisation Due to Worsening Renal Function
Description: Hospitalization due to worsening renal function (as per physician's decision) was defined as an overnight stay, or longer, in a hospital environment (emergency room, observation unit or in-patient care, or similar facility including admission to a day care facility) due to worsening renal function as the primary reason for hospitalization. Hazard ratio of Eplerenone versus placebo for first occurrence of the event was obtained from a Cox proportional hazards model.
Time Frame: Randomization up to the date when the last enrolled participant had been followed up for 1 year (up to 1744 days)
Population: Full analysis set included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 111 | 110
participants | 2 | 2
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.16 to 8.04]

16. Secondary Outcome: Number of Participants With First Occurrence of Hospitalization for Hyperkalemia
Description: Hospitalization due to hyperkalemia (as per physician's decision) was defined as an overnight stay, or longer, in a hospital environment (emergency room, observation unit or in-patient care, or similar facility including admission to a day care facility) due to hyperkalemia as the primary reason for hospitalization. Hazard ratio of Eplerenone versus placebo for first occurrence of the event was obtained from a Cox proportional hazards model.
Time Frame: Randomization up to the date when the last enrolled participant had been followed up for 1 year (up to 1744 days)
Population: Full analysis set included all randomized participants.
Measure: Number; unit: participants
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 111 | 110
participants | 0 | 0

17. Secondary Outcome: Change From Baseline in Plasma Concentration of Brain Natriuretic Peptide at Months 5, 9, 13, 17, 21, 25, 29, 33, 37, 42, 48 and Final Visit
Time Frame: Baseline, Months 5,9,13,17,21,25,29,33,37,42,48, Final Visit (up to Month 48)
Population: Full analysis set included all randomized participants. Here, 'n' signifies those participants who were evaluable at specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/ml)
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 111 | 110
picogram/milliliter (pg/ml)
  Baseline (n=111,110) | 469.29 (375.43) | 435.61 (391.49)
  Change at Month 5 (n=105,106) | -169.75 (424.40) | -36.36 (413.73)
  Change at Month 9 (n=99,104) | -208.54 (405.74) | -76.23 (442.47)
  Change at Month 13 (n=95,101) | -258.66 (395.05) | -93.99 (409.87)
  Change at Month 17 (n=81,82) | -242.92 (431.59) | -69.74 (535.05)
  Change at Month 21 (n=72,73) | -241.33 (429.24) | -57.31 (515.76)
  Change at Month 25 (n=63,63) | -249.76 (473.68) | -83.99 (506.79)
  Change at Month 29 (n=53,48) | -269.07 (502.78) | -95.33 (350.51)
  Change at Month 33 (n=45,40) | -228.84 (575.05) | -43.98 (500.78)
  Change at Month 37 (n=40,33) | -211.86 (597.30) | -73.73 (626.13)
  Change at Month 42 (n=30,26) | -155.65 (320.44) | -22.31 (689.26)
  Change at Month 48 (n=16,16) | -200.85 (357.51) | -122.33 (450.87)
  Change at Final Visit (n=109,110) | -149.75 (473.95) | -57.45 (509.85)
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; Change from baseline at Month 5 : Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -102.93, 95% CI 2-sided [-195.92 to -9.94], Standard Error of Mean 47.13
Statistical Analysis 2: Comparison: Eplerenone vs Placebo; Change from baseline at Month 9 :Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -95.77, 95% CI 2-sided [-184.51 to -7.04], Standard Error of Mean 44.54
Statistical Analysis 3: Comparison: Eplerenone vs Placebo; Change from baseline at Month 13 : Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -125.09, 95% CI 2-sided [-195.50 to -54.68], Standard Error of Mean 35.15
Statistical Analysis 4: Comparison: Eplerenone vs Placebo; Change from baseline at Month 17 :Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -31.94, 95% CI 2-sided [-232.77 to -31.11], Standard Error of Mean 51.12
Statistical Analysis 5: Comparison: Eplerenone vs Placebo; Change from baseline at Month 21 : Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -132.39, 95% CI 2-sided [-240.94 to -23.84], Standard Error of Mean 52.77
Statistical Analysis 6: Comparison: Eplerenone vs Placebo; Change from baseline at Month 25 :Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -117.18, 95% CI 2-sided [-221.49 to -12.87], Standard Error of Mean 51.76
Statistical Analysis 7: Comparison: Eplerenone vs Placebo; Change from baseline at Month 29 :Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -101.50, 95% CI 2-sided [-267.36 to 64.36], Standard Error of Mean 61.05
Statistical Analysis 8: Comparison: Eplerenone vs Placebo; Change from baseline at Month 33 : Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -110.78, 95% CI 2-sided [-307.49 to 85.93], Standard Error of Mean 92.42
Statistical Analysis 9: Comparison: Eplerenone vs Placebo; Change from baseline at Month 37 : Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -119.62, 95% CI 2-sided [-2137.82 to 1898.59], Standard Error of Mean 158.84
Statistical Analysis 10: Comparison: Eplerenone vs Placebo; Change from baseline at Month 42 : Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -144.60, 90% CI 2-sided [-2692.95 to 2403.76], Standard Error of Mean 200.56
Statistical Analysis 11: Comparison: Eplerenone vs Placebo; Change from baseline at Month 48 :Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -77.26, 95% CI 2-sided [-2131.88 to 1977.37], Standard Error of Mean 966.09
Statistical Analysis 12: Comparison: Eplerenone vs Placebo; Change from baseline at Month 13 : ANCOVA with treatment effect and covariates of the NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -102.30, 95% CI 2-sided [-172.61 to -32.00], Standard Error of Mean 35.67

18. Secondary Outcome: Change From Baseline in Plasma Concentration of Serum N-terminal Pro-Brain Natriuretic Peptide (NT-proBNP) at Months 5, 9, 13, 17, 21, 25, 29, 33, 37, 42, 48 and Final Visit
Time Frame: Baseline, Months 5, 9, 13, 17, 21 ,25, 29, 33, 37, 42, 48 and Final Visit (up to Month 48)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 111 | 110
pg/mL
  Baseline (n=111,110) | 2635.78 (2143.64) | 2354.31 (1874.30)
  Change at Month 5 (n=105,106) | -770.51 (2172.88) | -205.18 (1801.42)
  Change at Month 9 (n=99,104) | -884.76 (2265.57) | -425.47 (1883.54)
  Change at Month 13 (n=95,101) | -1066.86 (2088.51) | -452.02 (1878.98)
  Change at Month 17 (n=81,82) | -1126.96 (2384.14) | -109.59 (3380.42)
  Change at Month 21 (n=72,73) | -957.86 (2601.47) | -250.85 (2508.01)
  Change at Month 25 (n=63,63) | -453.57 (4894.51) | -128.02 (2627.01)
  Change at Month 29 (n=53,48) | -1013.83 (3167.91) | -187.08 (2524.52)
  Change at Month 33 (n=45,40) | -168.36 (5404.82) | 434.35 (5134.98)
  Change at Month 37 (n=40,33) | -9.64 (5188.24) | 171.21 (5081.43)
  Change at Month 42 (n=30,26) | -246.77 (4753.87) | 928.35 (6494.32)
  Change at Month 48 (n=16,16) | -970.71 (4833.60) | -450.69 (1487.78)
  Change at Final Visit (n=109,110) | -177.00 (3780.44) | 296.35 (3823.59)
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; Change from baseline at Month 5 :Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -364.65, 95% CI 2-sided [-1863.06 to 1133.76], Standard Error of Mean 763.83
Statistical Analysis 2: Comparison: Eplerenone vs Placebo; Change from baseline at Month 9 : Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -247.14, 95% CI 2-sided [-1642.43 to 1148.14], Standard Error of Mean 711.26
Statistical Analysis 3: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 17, analysis 3]; Test type: Superiority or Other; Least Square Mean Difference = -370.14, 95% CI 2-sided [-1742.51 to 1002.22], Standard Error of Mean 699.58
Statistical Analysis 4: Comparison: Eplerenone vs Placebo; Change from baseline at Month 17 : Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -664.09, 95% CI 2-sided [-141189.93 to 139861.75], Standard Error of Mean 11059.62
Statistical Analysis 5: Comparison: Eplerenone vs Placebo; Change from baseline at Month 21 :Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -414.99, 95% CI 2-sided [-39445.52 to 38615.54], Standard Error of Mean 3071.77
Statistical Analysis 6: Comparison: Eplerenone vs Placebo; Change from baseline at Month 25 : Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = 23.86, 95% CI 2-sided [-21649.89 to 21697.60], Standard Error of Mean 10794.85
Statistical Analysis 7: Comparison: Eplerenone vs Placebo; Change from baseline at Month 29 : Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -245.23, 95% CI 2-sided [-85358.69 to 84868.22], Standard Error of Mean 6698.57
Statistical Analysis 8: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 17, analysis 8]; Test type: Superiority or Other; Least Square Mean Difference = 170.49, 95% CI 2-sided [-21375.69 to 21716.66], Standard Error of Mean 10730.38
Statistical Analysis 9: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 17, analysis 9]; Test type: Superiority or Other; Least Square Mean Difference = -58.77, 95% CI 2-sided [-30160.25 to 30042.70], Standard Error of Mean 12765.30
Statistical Analysis 10: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 17, analysis 10]; Test type: Superiority or Other; Least Square Mean Difference = -212.25, 90% CI 2-sided [-22723.82 to 22299.33], Standard Error of Mean 11073.11
Statistical Analysis 11: Comparison: Eplerenone vs Placebo; Change from baseline at Month 48 : Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -80.16, 95% CI 2-sided [-146026.28 to 145865.96], Standard Error of Mean 11486.21
Statistical Analysis 12: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 17, analysis 12]; Test type: Superiority or Other; Least Square Mean Difference = -187.72, 95% CI 2-sided [-662.67 to 287.23], Standard Error of Mean 240.96

19. Secondary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF) at Months 5, 9, 13, 17, 21, 25, 29, 33, 37, 42, 48 and Final Visit
Description: LVEF was calculated based on end-diastolic volume measured by two-dimensional echocardiography.
Time Frame: Baseline, Months 5, 9, 13, 17, 21, 25, 29, 33, 37, 42, 48, Final Visit (up to Month 48)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: percentage of LVEF
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 111 | 110
percentage of LVEF
  Baseline (n=111,110) | 25.64 (4.95) | 26.64 (3.97)
  Change at Month 5 (n=105,106) | 5.98 (8.87) | 4.01 (7.59)
  Change at Month 9 (n=99,104) | 33.89 (10.64) | 31.37 (9.19)
  Change at Month 13 (n=94,101) | 9.62 (9.70) | 4.86 (10.13)
  Change at Month 17 (n=81,82) | 11.36 (11.45) | 5.50 (10.74)
  Change at Month 21 (n=72,73) | 12.73 (12.04) | 6.37 (11.88)
  Change at Month 25 (n=63,64) | 12.18 (12.18) | 6.60 (10.94)
  Change at Month 29 (n=53,48) | 11.95 (12.28) | 6.45 (12.83)
  Change at Month 33 (n=45,39) | 13.67 (13.94) | 5.20 (10.19)
  Change at Month 37 (n=40,33) | 13.34 (14.59) | 7.18 (10.49)
  Change at Month 42 (n=30,26) | 12.15 (14.38) | 5.13 (10.36)
  Change at Month 48 (n=16,16) | 10.18 (16.02) | 8.41 (11.51)
  Change at Final Visit (n=109,110) | 9.50 (12.03) | 5.99 (11.04)
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 1.71, 95% CI 2-sided [-0.55 to 3.96], Standard Error of Mean 1.14
Statistical Analysis 2: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 18, analysis 2]; Test type: Superiority or Other; Least Square Mean Difference = 2.74, 95% CI 2-sided [0.07 to 5.42], Standard Error of Mean 1.36
Statistical Analysis 3: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 17, analysis 3]; Test type: Superiority or Other; Least Square Mean Difference = 3.86, 95% CI 2-sided [1.11 to 6.60], Standard Error of Mean 1.39
Statistical Analysis 4: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 18, analysis 4]; Test type: Superiority or Other; Least Square Mean Difference = 4.86, 95% CI 2-sided [1.81 to 7.90], Standard Error of Mean 1.54
Statistical Analysis 5: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 17, analysis 5]; Test type: Superiority or Other; Least Square Mean Difference = 5.65, 95% CI 2-sided [2.36 to 8.94], Standard Error of Mean 1.67
Statistical Analysis 6: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 17, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = 3.44, 95% CI 2-sided [0.12 to 6.75], Standard Error of Mean 1.68
Statistical Analysis 7: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 18, analysis 7]; Test type: Superiority or Other; Least Square Mean Difference = 3.60, 95% CI 2-sided [-0.06 to 7.25], Standard Error of Mean 1.85
Statistical Analysis 8: Comparison: Eplerenone vs Placebo; Change from baseline at Month 33 :Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = 4.65, 95% CI 2-sided [0.86 to 8.44], Standard Error of Mean 1.92
Statistical Analysis 9: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 17, analysis 9]; Test type: Superiority or Other; Least Square Mean Difference = 3.85, 95% CI 2-sided [0.02 to 7.68], Standard Error of Mean 1.94
Statistical Analysis 10: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 17, analysis 10]; Test type: Superiority or Other; Least Square Mean Difference = 4.67, 90% CI 2-sided [0.08 to 9.25], Standard Error of Mean 2.31
Statistical Analysis 11: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 18, analysis 11]; Test type: Superiority or Other; Least Square Mean Difference = 4.13, 95% CI 2-sided [-1.82 to 10.07], Standard Error of Mean 2.98
Statistical Analysis 12: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 17, analysis 12]; Test type: Superiority or Other; Least Square Mean Difference = 3.18, 95% CI 2-sided [0.56 to 5.80], Standard Error of Mean 1.33

20. Secondary Outcome: Change From Baseline in Urine Albumin-to-Creatinine Ratio at Months 5, 9, 13, 17, 21, 25, 29, 33, 37, 42, 48 and Final Visit
Time Frame: Baseline, Months 5, 9, 13, 17, 21, 25, 29, 33, 37, 42, 48, Final Visit (up to Month 48)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: microgram per gram creatinine (mg/gCr)
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 111 | 110
microgram per gram creatinine (mg/gCr)
  Baseline (n=111,108) | 169.82 (787.32) | 154.93 (366.44)
  Change at Month 5 (n=104,103) | -21.14 (359.53) | 46.23 (377.56)
  Change at Month 9 (n=98,101) | -11.10 (249.68) | 23.79 (362.35)
  Change at Month 13 (n=94,98) | -41.56 (322.12) | -19.04 (253.57)
  Change at Month 17 (n=80,82) | -13.66 (247.48) | 79.28 (530.74)
  Change at Month 21 (n=72,73) | -63.65 (498.00) | 28.84 (431.48)
  Change at Month 25 (n=62,63) | 17.17 (489.08) | 30.08 (350.86)
  Change at Month 29 (n=50,47) | 18.51 (454.75) | -4.58 (504.53)
  Change at Month 33 (n=43,39) | -47.07 (506.66) | -3.38 (417.43)
  Change at Month 37 (n=39,33) | -80.21 (743.85) | 34.20 (393.95)
  Change at Month 42 (n=27,25) | -162.18 (921.61) | -29.95 (187.19)
  Change at Month 48 (n=16,16) | -303.19 (1211.28) | -41.03 (113.70)
  Change at Final Visit (n=109,110) | -29.30 (597.07) | -31.56 (271.71)
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; Change from baseline at Month 5: Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -61.53, 95% CI 2-sided [-186.44 to 63.37], Standard Error of Mean 59.75
Statistical Analysis 2: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 18, analysis 2]; Test type: Superiority or Other; Least Square Mean Difference = -24.94, 95% CI 2-sided [-131.27 to 81.39], Standard Error of Mean 54.20
Statistical Analysis 3: Comparison: Eplerenone vs Placebo; Change from baseline at Month 13 :Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -12.57, 95% CI 2-sided [-97.28 to 72.13], Standard Error of Mean 43.18
Statistical Analysis 4: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 17, analysis 4]; Test type: Superiority or Other; Least Square Mean Difference = -78.47, 95% CI 2-sided [-221.25 to 64.31], Standard Error of Mean 72.78
Statistical Analysis 5: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 17, analysis 5]; Test type: Superiority or Other; Least Square Mean Difference = -79.63, 95% CI 2-sided [-211.88 to 52.63], Standard Error of Mean 67.42
Statistical Analysis 6: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 18, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = 19.35, 95% CI 2-sided [-230.01 to 268.71], Standard Error of Mean 88.95
Statistical Analysis 7: Comparison: Eplerenone vs Placebo; Change from baseline at Month 29: Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -21.05, 95% CI 2-sided [-194.21 to 152.11], Standard Error of Mean 88.27
Statistical Analysis 8: Comparison: Eplerenone vs Placebo; Change from baseline at Month 33: Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -40.79, 95% CI 2-sided [-197.55 to 115.97], Standard Error of Mean 79.91
Statistical Analysis 9: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 17, analysis 9]; Test type: Superiority or Other; Least Square Mean Difference = -44.48, 95% CI 2-sided [-247.11 to 158.15], Standard Error of Mean 103.29
Statistical Analysis 10: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 17, analysis 10]; Test type: Superiority or Other; Least Square Mean Difference = -27.69, 90% CI 2-sided [-238.31 to 182.93], Standard Error of Mean 107.06
Statistical Analysis 11: Comparison: Eplerenone vs Placebo; Change from baseline at Month 48: Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -31.46, 95% CI 2-sided [-221.17 to 158.24], Standard Error of Mean 96.48
Statistical Analysis 12: Comparison: Eplerenone vs Placebo; Change from baseline at Month 13 :ANCOVA with treatment effect and covariates of the NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -2.04, 95% CI 2-sided [-58.91 to 54.83], Standard Error of Mean 28.85

21. Secondary Outcome: Number of Participants With Change From Baseline in New York Heart Association (NYHA) Classification at Weeks 1, 4, Months 2, 3, 4, 5, 9, 13, 17 21, 25, 29, 33, 37, 42, 48 and Final Visit
Description: NYHA: classified as 'class I' (participants with cardiac disease but without resulting limitations of physical activity), 'class II' (participants with cardiac disease resulting in slight limitation of physical activity), 'class III' (participants with cardiac disease resulting in marked limitation of physical activity), 'class IV' (participants with cardiac disease resulting in inability to carry on any physical activity without discomfort). Participants with change from baseline were classified as 'improved' (positive change), 'no change' or 'worsened' (negative change).
Time Frame: Baseline, Weeks 1, 4, Months 2, 3, 4, 5, 9, 13, 17, 21, 25, 29, 33, 37, 42, 48 and Final Visit (up to Month 48)
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 111 | 110
participants
  Week 1 (n=111, 110) : Improved | 4 | 2
  Week 1 (n=111, 110) : Unchanged | 107 | 107
  Week 1 (n=111, 110) : Worse | 0 | 1
  Week 4 (n=111, 108) : Improved | 10 | 14
  Week 4 (n=111, 108) : Unchanged | 101 | 92
  Week 4 (n=111, 108) : Worse | 0 | 2
  Month 2 (n=109, 109) : Improved | 15 | 14
  Month 2 (n=109, 109) : Unchanged | 94 | 95
  Month 2 (n=109, 109) : Worse | 0 | 0
  Month 3 (n=106, 107) : Improved | 18 | 16
  Month 3 (n=106, 107) : Unchanged | 88 | 91
  Month 3 (n=106, 107) : Worse | 0 | 0
  Month 4 (n=106, 106) : Improved | 22 | 20
  Month 4 (n=106, 106) : Unchanged | 82 | 86
  Month 4 (n=106, 106) : Worse | 2 | 0
  Month 5 (n=104, 106) : Improved | 24 | 22
  Month 5 (n=104, 106) : Unchanged | 76 | 83
  Month 5 (n=104, 106) : Worse | 4 | 1
  Month 9 (n=99, 105) : Improved | 27 | 20
  Month 9 (n=99, 105) : Unchanged | 71 | 81
  Month 9 (n=99, 105) : Worse | 1 | 4
  Month 13 (n=94, 102) : Improved | 31 | 19
  Month 13 (n=94, 102) : Unchanged | 62 | 82
  Month 13 (n=94, 102) : Worse | 1 | 1
  Month 17 (n=81, 82) : Improved | 25 | 18
  Month 17 (n=81, 82) : Unchanged | 55 | 61
  Month 17 (n=81, 82) : Worse | 1 | 3
  Month 21 (n=72, 73) : Improved | 21 | 19
  Month 21 (n=72, 73) : Unchanged | 50 | 51
  Month 21 (n=72, 73) : Worse | 1 | 3
  Month 25 (n=63, 64) : Improved | 23 | 14
  Month 25 (n=63, 64) : Unchanged | 38 | 48
  Month 25 (n=63, 64) : Worse | 2 | 2
  Month 29 (n=53, 48) : Improved | 17 | 12
  Month 29 (n=53, 48) : Unchanged | 36 | 35
  Month 29 (n=53, 48) : Worse | 0 | 1
  Month 33 (n=46, 39) : Improved | 14 | 10
  Month 33 (n=46, 39) : Unchanged | 31 | 27
  Month 33 (n=46, 39) : Worse | 1 | 2
  Month 37 (n=40, 33) : Improved | 12 | 10
  Month 37 (n=40, 33) : Unchanged | 28 | 22
  Month 37 (n=40, 33) : Worse | 0 | 1
  Month 42 (n=30, 26) : Improved | 7 | 7
  Month 42 (n=30, 26) : Unchanged | 23 | 18
  Month 42 (n=30, 26) : Worse | 0 | 1
  Month 48 (n=16, 16) : Improved | 2 | 6
  Month 48 (n=16, 16) : Unchanged | 14 | 9
  Month 48 (n=16, 16) : Worse | 0 | 1
  Final Visit (n=111, 110) : Improved | 25 | 26
  Final Visit (n=111, 110) : Unchanged | 80 | 80
  Final Visit (n=111, 110) : Worse | 6 | 4

22. Secondary Outcome: Change From Baseline in Specific Activity Scale (SAS) Score at Week 4, Months 2, 3, 4, 5, 9, 13, 17 21, 25, 29, 33, 37, 42, 48 and Final Visit
Description: Specific activity scale was estimated by pre-specified questionnaire (for different activities) to assess the exercise capability of the participants. Answers provided by participants were transformed in terms of number of metabolic equivalents (METs).1 MET was defined as the amount of oxygen consumed while sitting at rest and is equal to 3.5 ml oxygen per kg body weight* minute. Scale ranged from 1 (less than (<) 2 METs) = lowest level of exercise tolerance to 6 (>=8METs) = highest level of tolerance and higher score indicated more tolerance.
Time Frame: Baseline, Week 4, Months 5, 9, 13, 17, 21, 25, 29, 33, 37, 42, 48, Final Visit (up to Month 48)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: metabolic equivalents (METs)
Arm/Group | Eplerenone | Placebo
Number analyzed (Participants) | 111 | 110
metabolic equivalents (METs)
  Baseline (n=111,110) | 4.85 (1.51) | 4.89 (1.54)
  Change at Week 4 (n= 111,108) | 0.15 (0.79) | 0.27 (1.08)
  Change at Month 5 (n=104,106) | 0.46 (1.15) | 0.33 (1.19)
  Change at Month 9 (n=99,104) | 0.41 (1.16) | 0.37 (1.39)
  Change at Month 13 (n=94,102) | 0.52 (1.18) | 0.44 (1.45)
  Change at Month 17 (n=81,82) | 0.46 (1.38) | 0.47 (1.81)
  Change at Month 21 (n=72,73) | 0.34 (1.33) | 0.59 (1.64)
  Change at Month 25 (n=63,63) | 0.48 (1.08) | 0.63 (1.72)
  Change at Month 29 (n=53,48) | 0.42 (1.14) | 0.65 (1.56)
  Change at Month 33 (n=46,40) | 0.37 (1.28) | 0.51 (1.80)
  Change at Month 37 (n=40,33) | 0.53 (1.47) | 0.68 (1.39)
  Change at Month 42 (n=30,26) | 0.39 (1.70) | 0.47 (1.83)
  Change at Month 48 (n=16,16) | -0.13 (1.57) | 0.64 (1.59)
  Change at Final Visit (n=111,110) | 0.14 (1.56) | 0.25 (1.65)
Statistical Analysis 1: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 0.08, 95% CI 2-sided [-0.21 to 0.37], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 17, analysis 2]; Test type: Superiority or Other; Least Square Mean Difference = -0.02, 95% CI 2-sided [-0.34 to 0.30], Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: Eplerenone vs Placebo; Change from baseline at Month 13: Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = 0.06, 95% CI 2-sided [-0.27 to 0.39], Standard Error of Mean 0.17
Statistical Analysis 4: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 18, analysis 4]; Test type: Superiority or Other; Least Square Mean Difference = 0.02, 95% CI 2-sided [-0.41 to 0.45], Standard Error of Mean 0.22
Statistical Analysis 5: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 17, analysis 5]; Test type: Superiority or Other; Least Square Mean Difference = -0.16, 95% CI 2-sided [-0.56 to 0.24], Standard Error of Mean 0.20
Statistical Analysis 6: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 18, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = -0.15, 95% CI 2-sided [-0.55 to 0.25], Standard Error of Mean 0.20
Statistical Analysis 7: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 18, analysis 7]; Test type: Superiority or Other; Least Square Mean Difference = -0.09, 95% CI 2-sided [-0.49 to 0.31], Standard Error of Mean 0.20
Statistical Analysis 8: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 17, analysis 8]; Test type: Superiority or Other; Least Square Mean Difference = -0.07, 95% CI 2-sided [-0.57 to 0.44], Standard Error of Mean 0.26
Statistical Analysis 9: Comparison: Eplerenone vs Placebo; Change from baseline at Month 37 :Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = 0.02, 95% CI 2-sided [-0.50 to 0.54], Standard Error of Mean 0.26
Statistical Analysis 10: Comparison: Eplerenone vs Placebo; Change from baseline at Month 42 :Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = 0.20, 90% CI 2-sided [-0.44 to 0.83], Standard Error of Mean 0.32
Statistical Analysis 11: Comparison: Eplerenone vs Placebo; [analysis description as in outcome 18, analysis 11]; Test type: Superiority or Other; Least Square Mean Difference = 0.13, 95% CI 2-sided [-0.63 to 0.89], Standard Error of Mean 0.38
Statistical Analysis 12: Comparison: Eplerenone vs Placebo; Change from baseline at Week 4 : Mixed effect model of repeated measurements with covariates of the treatment, Week, interaction between treatment and week, baseline NYHA cohort (II, III/IV), baseline eGFR (30-<50 ml/min/1.73 m^2, >=50 ml/min/1.73 m^2) and baseline value; Test type: Superiority or Other; Least Square Mean Difference = -0.13, 95% CI 2-sided [-0.36 to 0.11], Standard Error of Mean 0.12

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event and an serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non serious event during the study.
Arm/Group | Eplerenone | Placebo
Serious Adverse Events (participants affected / at risk) | 52/111 | 65/110
Other Adverse Events (participants affected / at risk) | 89/111 | 87/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eplerenone (N=111) | Placebo (N=110)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 0
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 2 | 4
Angina unstable (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2
Atrial flutter (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 27 | 31
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 2
Cardiac sarcoidosis (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 2 | 2
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 5 | 3
Cataract (Eye disorders) | 2 | 3
Retinal detachment (Eye disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Protein-losing gastroenteropathy (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 1 | 2
Sudden death (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 3
Appendicitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 2
Disseminated tuberculosis (Infections and infestations) | 0 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 5
Pneumonia bacterial (Infections and infestations) | 0 | 2
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 0
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 | 1
Blood pressure decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 3 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cervical myelopathy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Spondylitic myelopathy (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 1
Renal impairment (Renal and urinary disorders) | 0 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 2
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Eplerenone (N=111) | Placebo (N=110)
Anaemia (Blood and lymphatic system disorders) | 7 | 6
Cardiac failure (Cardiac disorders) | 21 | 32
Chronic gastritis (Gastrointestinal disorders) | 6 | 3
Constipation (Gastrointestinal disorders) | 8 | 18
Diarrhoea (Gastrointestinal disorders) | 7 | 10
Haemorrhoids (Gastrointestinal disorders) | 2 | 6
Hepatic function abnormal (Hepatobiliary disorders) | 4 | 7
Bronchitis (Infections and infestations) | 6 | 8
Conjunctivitis (Infections and infestations) | 7 | 5
Nasopharyngitis (Infections and infestations) | 37 | 40
Upper respiratory tract infection (Infections and infestations) | 5 | 6
Contusion (Injury, poisoning and procedural complications) | 12 | 5
Fall (Injury, poisoning and procedural complications) | 20 | 20
Blood pressure decreased (Investigations) | 6 | 4
Dehydration (Metabolism and nutrition disorders) | 10 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 7 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 11 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 3
Dizziness (Nervous system disorders) | 8 | 5
Renal impairment (Renal and urinary disorders) | 5 | 7
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0/26 | 1/19 — As the event is gender specific, only female participants were evaluated.
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 8
Eczema (Skin and subcutaneous tissue disorders) | 4 | 6
Hypertension (Vascular disorders) | 9 | 3
Hypotension (Vascular disorders) | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.